# Statistical Analysis Plan with Amendment 02

A Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Multiple-Site Clinical Study to Evaluate the Therapeutic Equivalence and Safety of Ivermectin Lotion 0.5% (Actavis Laboratories UT, Inc.) to SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC) in the Treatment of Human Head Lice Infestation

**Study Number 71691702** 

NCT03301649

Statistical Analysis Plan with Amendment 02 Approval Date: 12 January 2018

A Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Multiple-Site Clinical Study to Evaluate the Therapeutic Equivalence and Safety of Ivermectin Lotion 0.5% (Actavis Laboratories UT, Inc.) to SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC) in the Treatment of Human Head Lice Infestation

Protocol Number: 71691702 71691702

# **Sponsor:**

Actavis LLC 400 Interpace Parkway Morris Corporate Center III Parsippany, NJ 07054



January 12, 2018

Draft Version 2.0

Protocol / Study No. 71691702

## **SAP FINAL VERSION APPROVALS**

A Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Multiple-Site Clinical Study to Evaluate the Therapeutic Equivalence and Safety of Ivermectin Lotion 0.5% (Actavis Laboratories UT, Inc.) to SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC) in the Treatment of Human Head Lice Infestation

| Written By: | |
|--------------|-------|
| Signature: | Date: |
| Reviewed By: | |
| Signature: | Date: |
| Approved By: | |
| Signature: | Date: |
| Actavis LLC | |

01/12/2017 ■ Actavis LLC■ 

**Ivermectin Lotion 0.5%** 

Protocol / Study No. 71691702

# **Revision History**

| VERSION | DATE | DESCRIPTION OF REVISIONS | REVISED BY |
|-----------|-------------------|-----------------------------|------------|
| Draft 1.0 | December 06, 2017 | New Document | |
| Draft 2.0 | January 12, 2018 | Incorporate client comments | |

#### **Ivermectin Lotion 0.5%**

Protocol / Study No. 71691702

# List of Abbreviations and Definition of Terms

ADaM Analysis Data Model

AE Adverse Event

ANOVA Analysis of Variance

C Celsius

CDISC Clinical Data Interchange Standards Consortium

CMH Cochran-Mantel-Haenszel

CRF Case Report Form

CRO Contract Research Organization

EOS End of Study Fahrenheit

FDA Food and Drug Administration GLM Generalized Linear Model

Hg Mercury

ICF Informed Consent Form

ICH International Conference on Harmonisation

IWRS Interactive Web Response System LOCF Last Observation Carried Forward

MedDRA Medical Dictionary for Regulatory Activities

mITT modified Intent-to-Treat Population

OGD Office of Generic Drugs
PP Per-Protocol Population
RLD Reference Listed Drug
SAE Serious Adverse Event
SAP Statistical Analysis Plan
SAS Statistical Analysis System

SD Standard Deviation

SDTM Study Data Tabulation Model

**Ivermectin Lotion 0.5%** 

Protocol / Study No. 71691702

# TABLE OF CONTENTS

| 1. INTRODUCTION | 7 |
|---|---|
| 2. OBJECTIVES | |
| 3. OVERALL STUDY DESIGN | 7 |
| 4. RANDOMIZATION AND BLINDING | 11 |
| 5. SAMPLE SIZE | |
| 6. ANALYSIS POPULATION | 12 |
| 7. EFFICACY ENDPOINTS | 13 |
| 8. STATISTICAL ANALYSIS METHODS | 13 |
| 8.1 Baseline Characteristics | 14 |
| 8.1.1 Baseline Comparability | 14 |
| 8.1.2 Medical History | |
| 8.1.3 Concomitant Medications | 14 |
| 8.1.4 Pregnancy Test | 15 |
| 8.2 Efficacy Analyses | 15 |
| 8.2.1 Primary and Secondary Endpoint Analysis | 15 |
| 8.2.2 Treatment-by-Site Interaction and Pooling of Clinical Sites | |
| 8.3 Safety Analysis | 17 |
| 8.3.1 Adverse Events | 17 |
| 8.3.2 Application Site Reactions | 17 |
| 8.3.3 Vital Signs | 18 |
| 8.4 Multiple Comparisons | 18 |
| 8.5 Methods for Handling Missing Data | 18 |
| 8.6 Interim Analyses | 18 |
| 9. TABLE, LISTING AND FIGURE SHELLS | 19 |
| T16.1.9.1 Summary of Discontinued Patients | 21 |
| T16.1.9.2 Summary of Protocol Deviations | 22 |
| T16.1.9.3.1 Summary of Patients Excluded from Efficacy Analysis | 23 |
| T16.1.9.3.2 Summary of Patients Included in Analysis Population by Study Center | 25 |
| T16.1.9.4 Summary of Demographic Data and Baseline Characteristics (Safety Popula | ation) |
| T16.1.9.5 Summary of Demographic Data and Baseline Characteristics (modified Inter | nt-to-Trea |
| Population) | 28 |
| T16.1.9.6 Summary of Demographic Data and Baseline Characteristics (Per-Protocol | |
| Population) | |
| T16.1.9.7.1 Summary of Analysis Results of Primary Efficacy Endpoint | 29 |
| T16.1.9.7.2 Sensitivity Analysis Results of Primary Efficacy EndpointError! Bookma | rk not |
| defined. | |
| T16.1.9.7.3 Sensitivity Analysis Results of Primary Efficacy EndpointError! Bookma | ırk not |
| defined. | |

# **Ivermectin Lotion 0.5%**

# Protocol / Study No. 71691702

| T16.1.9.8 Summary of Analysis Results of Secondary Efficacy Endpoint | |
|---|---|
| T16.1.9.9 Overall Summary of Adverse Events (Safety Population) | |
| T16.1.9.10 Summary of Frequency of All Adverse Events by Body System (Safety Population | on) |
| 32 | ĺ |
| T16.1.9.11 Summary of Frequency of All Adverse Events by Severity (Safety Population)33 | |
| T16.1.9.12 Summary of Frequency of All Adverse Events by Relationship (Safety Population | n) |
| 34 | |
| T16.1.9.13 Summary of Frequency of Serious Adverse Events (Safety Population) 35 | |
| T16.1.9.14 Summary of Frequency of Application Site Reaction (Safety Population) 36 | |
| T16.1.9.15 Summary of Vital Signs (Safety Population) | |
| T16.1.9.16 Summary of Frequence of Patients who are Treatment Failures at Visit 2 and Visit | t 3 |
| (Safety Population)38 | |
| T16.1.9.17 Summary of Fequency of Patients with Re-Infestation (Safety Population) 39 | |
| L16.2.1 Listing of Discontinued Patients | |
| L16.2.2 Listing of Protocol Deviations | |
| L16.2.3.1 Listing of Patients Excluded from the Per-Protocol Population | |
| L16.2.3.2 Lisitng of Patients Excluded from the Modified Intent-to-Treat Population 43 | |
| L16.2.4.1 Listing of Demographic Data | |
| L16.2.4.2 Listing of Medical History | |
| L16.2.4.3 Listing of Concomitant Medications | |
| L16.2.5 Listing of Visit Date Information | |
| L16.2.6 Listing of Louse Examination Results | |
| L16.2.7.1 Listing of Adverse Events by Treatment Group | |
| L16.2.7.2 Listing of Application Site Reactions | |
| L16.2.8.1 Listing of Pregnancy Test Results | |
| L16.2.8.2 Listing of Vital Signs | |

#### **Ivermectin Lotion 0.5%**

Protocol / Study No. 71691702

#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the final Clinical Study Protocol 71691702 Rev. 0 dated 06/21/2017. The SAP provides details on the planned statistical methodology for the analysis of the study data. The SAP also outlines the statistical programming specifications for the tables, listings and figures.

This SAP describes the study endpoints, derived variables, anticipated data transformations and manipulations, and other details of the analyses not provided in the study protocol. This SAP therefore outlines in detail all other aspects pertaining to the planned analyses and presentations for this study.

The following documents were reviewed in preparation of this SAP:

- Final Clinical Study Protocol 71691702 Rev.0 dated 06/21/2017
- Final eCRF Version 1.0 for Study No. 71691702

The reader of this SAP is encouraged to also read the clinical protocol for details on the conduct of this study, and the operational aspects of clinical assessments and timing for completing a patient in this study.

#### 2. OBJECTIVES

The objectives of this study are to:

- 1. Evaluate the therapeutic equivalence of the Test formulation, Ivermectin Lotion 0.5% (Actavis Laboratories UT, Inc.) to the Reference product, SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC) in the treatment of active head lice infestation.
- 2. Demonstrate the superiority of the Test and Reference (active) treatments over Placebo treatment in patients with active head lice infestation.
- 3. Compare the safety of Test, Reference and Placebo treatments in patients with active head lice infestation.

#### 3. OVERALL STUDY DESIGN

This randomized, double-blind, placebo-controlled, parallel-design, multiple-site clinical study has been designed to evaluate the efficacy and safety of a generic Ivermectin Lotion 0.5% (Actavis Laboratories UT, Inc.) compared to the Food and Drug Administration (FDA) Reference Listed Drug (RLD) SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals,

#### **Ivermectin Lotion 0.5%**

Protocol / Study No. 71691702

LLC) in patients with active head lice infestation. Additionally, both the Test and Reference (i.e., the RLD) treatments will be tested for superiority to a Placebo.

Before any study-specific procedures are performed, all patients will read and sign the IRB-approved informed consent form (ICF). In addition, patients who are considered minors in the state the study is being conducted (< 18 years of age in most states), must have a signed parental/guardian ICF, indicating approval to participate, as well as a signed assent to participate form, as appropriate. Patients 11-17 years of age will read and sign an IRB-approved assent form and patients 6-10 years of age will provide verbal assent. Patients 6 months-5 years of age will be exempt from providing assent based on the child's comprehension and cognitive skills.

Males and females, 6 months of age and older with an active head lice infestation will be randomized to one of the three study products as follows:

- **Test**: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)
- **Reference**: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)
- Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

Patients, will be instructed to administer a single application of the study product to the hair on the day of or the day after enrollment into the study, leave the study product on the hair and scalp for 10 minutes, and then rinse off with warm water. Patients and infested household members will be instructed to apply the study product at home. The day of dosing will be considered Day 1.

Patients will attend the following four scheduled clinics visits:

- Visit 1 (Day -1 to 1): Screening/Baseline
- Visit 2 (Day 2): Interim Visit
- Visit 3 (Day  $8 \pm 2$ ): Interim Visit
- Visit 4 (Day  $15 \pm 2$ ): End of Study

At Visit 2 (Day 2), enrolled will return the study product to the clinic. Visit 2 must occur the day after dosing.

At

Visits 2, 3, and 4, patients will be examined for the presence of live head lice (i.e., live adults

01/12/2017 ■ Actavis LLC■ 

# **Ivermectin Lotion 0.5%**

Protocol / Study No. 71691702

and/or nymphs). Louse examination should be conducted for 15 minutes or longer, unless any live lice are detected in less time. Duration of examination should be recorded.

Unscheduled visits will be allowed as deemed necessary by the Investigator or Sponsor to ensure patient safety or to perform other study-related procedures.

At Visit 2, patients will be questioned about any ocular discomfort associated with the study product. Also at Visits 2, 3, and 4, patients will be questioned about any adverse events (AEs), application site reactions (Appendix A), and any new concomitant medication use.

#### **Definitions**

- Non-index patient: Any household member who has agreed to participate in the study but is not the youngest member of the household.
- Index patient: The youngest household member who is randomized into the study.

Therapeutic equivalence will be assessed by evaluating the proportion of index patients in each treatment group who are considered a Treatment Success on Day  $15 \pm 2$ . Treatment Success is defined as the absence of live lice. The proportion of all patients (i.e., index + non-index) who are considered a Treatment Success on Day  $15 \pm 2$  will be evaluated as a secondary endpoint. The analysis of superiority will compare both active treatment groups to the Placebo group for the same primary and secondary endpoints.

# **Ivermectin Lotion 0.5%**

Protocol / Study No. 71691702

# **Study Schematic**

| PROCEDURE | VISIT 1 (Day -1 to 1)* Screening/Baseline | VISIT 2<br>(Day 2) <sup>†</sup><br>Interim<br>Visit | VISIT 3 (Day 8 ± 2 Days) Interim Visit | VISIT 4 (Day 15 ± 2 Days) End of Study |
|---|---|---|---|---|
| Informed | X | | | |
| Consent/Assent | | | | |
| Medical History and | X | | | |
| Demographics | | | | |
| Concomitant | X | X | X | X |
| Medication | | | | |
| Adverse Events | X | X | X | X |
| Vital Signs | X | X | X | X |
| Pregnancy Test <sup>‡</sup> | X | X | X | X |
| Louse Examination | X | X | X | X |
| Inclusion/Exclusion | X | | | |
| Application Site | X | X | X | X |
| Reactions | | | | |
| Ocular Irritation | | X | | |
| Assessment | | | | |
| Dispense Study | X | | | |
| Product | | | | |
| Collect Study Product | | X | | |
| Provide Patient Diary | X | X | X | |
| Collect and Review<br>Patient Diary | | X | X | X |

<sup>\*</sup>Study product will be administered on Day 1.

<sup>†</sup>Visit 2 must occur the day after patient dosing.

<sup>‡</sup>For females of childbearing potential

Protocol / Study No. 71691702

#### 4. RANDOMIZATION AND BLINDING

The study product will be randomized, packaged and blinded by an independent packaging company (Actavis, SLC site). The randomization will be pre-planned according to a computer-generated randomization schedule. All enrolled members of a household will be randomized to the same treatment arm.

Using Interactive Web Response Technology System (IWRS), all eligible and non-eligible patients who are consented and screened into the study will be assigned a patient number. The patient number is assigned after a patient is consented. It is the only identifier for screened patients.

The system will also assign a study product kit number (based on the randomization schedule created by an

also assign a study product kit number (based on the randomization schedule created by an independent biostatistician). The study product kit number is the identifying number listed on the study product dispensed to eligible patients. The study product kit number is a five-digit number. This will be the identifier used for randomized patients (i.e., randomization number). Both the patient number and randomization number will be entered into the patient's eCRF. At the end of the study, after all the clinical data have been entered and the study database has been locked, a copy of the randomization schedule will be sent to the statistician.

The Investigator, staff at the study site, study monitors, and data analysis/management personnel will be blinded to the patient assignment.

#### 5. SAMPLE SIZE

For the primary endpoint analysis (proportion of index patients in the PP population who are considered to be a Treatment Success on Day  $15 \pm 2$ ), sample size is estimated for therapeutic equivalence of the Test to the Reference product and superiority of each of the active treatments groups over Placebo. The sample size estimations are based on data reported in the product label for SKLICE® (ivermectin) Lotion, 0.5%.



# **Ivermectin Lotion 0.5%**

Protocol / Study No. 71691702



# **6. ANALYSIS POPULATION**

# **Per-Protocol Population (PPP)**

The PP population will include all randomized patients who:

- Meet all inclusion and exclusion criteria.

- Have no significant protocol deviations.
- Apply the study product as instructed on Day 1.



#### **Ivermectin Lotion 0.5%**

Protocol / Study No. 71691702

# **Modified Intent-to-Treat Population (mITT)**

The mITT population will include all randomized patients who meet all inclusion/exclusion criteria, apply the study product as instructed, and return for at least one post-baseline evaluation visit.

# **Safety Population**

The Safety population will include all patients who are randomized and received study product.

#### 7. EFFICACY ENDPOINTS

## **Primary Efficacy Endpoint**

The primary efficacy endpoint is the proportion of index patients in each treatment group who are considered a Treatment Success on Day  $15 \pm 2$ . Treatment Success is defined as the absence of live lice.

## **Secondary Efficacy Variable**

The secondary efficacy endpoint is the proportion of all randomized patients (i.e., index + non-index) who are considered a Treatment Success on Day  $15 \pm 2$ . Treatment Success is defined as the absence of live lice.

#### 8. STATISTICAL ANALYSIS METHODS

If not otherwise specified, statistical significance is defined as p < 0.05 and is two-tailed. Data will be summarized with respect to demographic and baseline characteristics, efficacy variables and safety variables.

For categorical variables, the number and percent of each category within a parameter will be calculated for non-missing data. For continuous variables, statistics will include number of observations, mean, standard deviation, median, minimum and maximum values.

All statistical analyses will be conducted using SAS®, Version 9.4 or higher. Datasets will be prepared using headings from Clinical Data Interchange Consortium (CDISC) Study Data Tabulation Model (SDTM) implementation for human clinical trials and ADaM (Analysis Dataset Model). ADaM datasets will include but not limited to ADSL, ADEFF, ADAE, ADVS, ADCM and ADMH.

#### **Ivermectin Lotion 0.5%**

Protocol / Study No. 71691702

#### 8.1 Baseline Characteristics

#### **8.1.1** Baseline Comparability

Baseline characteristics will be evaluated separately for the PP, mITT and Safety populations.

Demographic information collected at baseline includes the following:

- Age (years)
- Gender (Male/Female)
- Ethnicity (Hispanic/non Hispanic)
- Race (White, Black/African American, Native Hawaiian or Other Pacific Islander, Asian, American Indian or Alaska Native, Other)
- Number of live lice

Summary tables by treatment group will be presented. Continuous variables will be summarized using descriptive statistics (number of observations, median, minimum, maximum, mean and standard deviation). Categorical variables will be summarized using frequencies and percentage. Baseline treatment comparisons will be presented using Chi-Square test for the categorical variables, and Analysis of Variance (ANOVA) for the continuous variables.

All data will be listed by treatment and patient.

## **8.1.2** Medical History

At Visit 1, each patient will be required to provide basic demographic information: date of birth, gender, ethnicity and race. Patients will also be questioned about medical history, including acute and chronic medical history and medical history relevant to their head lice.

Medical history data will be listed by treatment and patient.

#### **8.1.3 Concomitant Medications**

At Visit 1, patients will be questioned about current and previous medication use over the last four weeks. At all subsequent visits, patients will be questioned about ongoing or new concomitant medication use.

All prior and concomitant medications taken since screening until the end of the study will be listed by treatment and patient.

# 8.1.4 Pregnancy Test

All females of childbearing potential will have a urine pregnancy test performed at each visit.

Pregnancy test results will be listed by treatment and patient.

# **8.2 Efficacy Analyses**

## 8.2.1 Primary and Secondary Endpoint Analysis

## **Therapeutic Bioequivalence Analysis**

The primary measure of therapeutic equivalence will be evaluated using the Per-Protocol population.

Based on the usual method used in OGD for binary outcomes, the 90% confidence interval for the difference in success proportions between test and reference treatment should be contained within [-0.20, +0.20] in order to establish equivalence.

The compound hypothesis to be tested is:

$$H_0: P_T - P_R \le -.20 \text{ or } P_T - P_R \ge .20 \text{ versus}$$

$$H_A : -.20 < P_T - P_R < .20$$

where  $P_{\tau}$  = success rate of test treatment

 $P_{\mathbb{R}}$  = success rate of reference treatment.

Let

 $n_T$  = sample size of test treatment group

 $cn_{\tau}$  = number of subjects considered as Treatment Success in test treatment group

 $n_{\mathbb{R}}$  = sample size of reference treatment group

 $cn_R$  = number of subjects considered as Treatment Success in reference treatment group

$$\hat{P}_T = c n_T / n_T$$
  $\hat{P}_R = c n_R / n_R$ , and

$$se = (\widehat{P}_T (1 - \widehat{P}_T)/n_T + (\widehat{P}_R (1 - \widehat{P}_R)/n_R)^{1/2})$$

The 90% confidence interval for the difference in proportions between test and reference will be calculated as follows:

#### **Ivermectin Lotion 0.5%**

Protocol / Study No. 71691702

$$L = (\hat{P}_T - \hat{P}_R) - 1.645 \text{ se}$$

$$U = (\hat{P}_T - \hat{P}_R) + 1.645 \text{ se}$$

If the 90% confidence interval for the absolute difference between the proportion of patients who are considered a Treatment Success in the Test and Reference groups is contained within the range [-20%, +20%] then therapeutic equivalence of the Test product to the Reference product will be considered to have been demonstrated.

The same statistical approach will be conducted for analysis of the secondary endpoint in the PP population.

To declare therapeutic equivalence of the Test product to the Reference product, therapeutic equivalence must be demonstrated for only the primary endpoint in the PP population.

# **Superiority to Placebo Analysis**

Superiority of the Test and Reference products against the Placebo for the primary endpoint will be tested at the 5% significance level (p < 0.05; two-sided, CMH test, stratified by clinical site) in the mITT population using last observation carried forward (LOCF). If the proportions of patients who are considered a Treatment Success in the Test and Reference groups are numerically and statistically superior to that of the Placebo (p < 0.05; using two-sided, CMH test stratified by clinical site), then superiority of the Test and Reference products over Placebo will be concluded.

The same statistical approach will be conducted for analysis of the secondary endpoint in the mITT population.

To declare superiority of the Test and Reference products over Placebo, their superiority must be demonstrated for only the primary endpoint in the mITT population.

# 8.2.2 Treatment-by-Site Interaction and Pooling of Clinical Sites

As this is a multiple-site study, the interaction of treatment-by-site may be evaluated for the primary efficacy endpoint in the PP population (for equivalence testing). The treatment-by-site interaction will be evaluated by the Breslow-Day test for homogeneity of the odds ratio at the 5% significance level (p < 0.05). A site(s) with a low enrollment rate(s) may be pooled with its geographically closest site, so as to avoid bias in the estimation of a treatment-by-site interaction effect. The pooling will be done for low enrolling sites that account for less than 4-7% of the total number of patients in the PP population at the site with the highest enrolling rate in the PP population. If the treatment-by-site interaction term is found to be statistically significant (p < 0.05) then the interaction term will also be assessed for clinical relevance before pooling the data

#### **Ivermectin Lotion 0.5%**

Protocol / Study No. 71691702

across sites. This will include examination of Treatment Success rates at each site where sample sizes per treatment may be influential in the assessment of the interaction.

# 8.3 Safety Analysis

All safety analyses will be based on the Safety Population.

#### **8.3.1** Adverse Events

All the adverse events (AEs) reported throughout the study will be coded and classified according to the MedDRA (Medical Dictionary for Regulatory Activities) coding dictionary (Version 20.0 or higher). Each adverse event is to be evaluated for date of start and end, seriousness, severity, causal relationship with the study drugs, action taken and outcome.

The total number and percentage of patients with at least one AEs, discontinued study drug due to AEs, AE severity and AEs related to investigational product, serious AEs and death will be summarized by treatment groups.

A summary table of the number and percent of patients with AEs by system organ class, preferred term, and treatment group will be presented. Each patient will be counted only once within each preferred term.

A frequency summary table of the number of AEs by system organ class, preferred term, severity, and treatment group will be presented. Severity will be classified as "Mild", "Moderate", or "Severe".

Similarly, a frequency summary table of the number of AEs by system organ class, preferred term, and relationship to a study drug, and treatment group will be presented. Relationship to a study drug will be classified as "Related" or "Not Related".

Adverse event frequencies will be compared between treatments using Fisher's exact test. If the overall Fisher's test is statistically significant, a pairwise test will be conducted for Test and Reference to determine if the difference in AEs is related to the active product.

#### **8.3.2** Application Site Reactions

The following application site reactions will be evaluated at each visit based on the scale provided below:

Signs and Symptoms:

Erythema

Pyoderma

## **Ivermectin Lotion 0.5%**

Protocol / Study No. 71691702

Excoriation

Pain

**Pruritus** 

Edema

Grading Scale:

Absent 0

Mild 1 (slight, barely perceptible)

Moderate 2 (distinct presence) Severe 3 (marked, intense)

Application site reactions and ocular discomfort will be compared descriptively among treatment groups. A frequency summary table comparing the application site reactions for each treatment group will be presented by visit.

# 8.3.3 Vital Signs

Vital signs will be recorded (pulse, blood pressure, temperature and respiration rate) at each visit.

Descriptive summaries (number of observations, mean, standard deviation, minimum, median and maximum) will be provided by treatment and visit.

All data will be listed by treatment and patient.

## 8.4 Multiple Comparisons

No multiple comparison adjustment will be made in this study.

# 8.5 Methods for Handling Missing Data

For demographic and baseline characteristics, each variable will be analyzed using all available data. Patients with missing data will be excluded only from analyses for which data are not available.

## 8.6 Interim Analyses

There is no interim analysis planned in this study.

**Ivermectin Lotion 0.5%** 

Protocol / Study No. 71691702

# 9. TABLE, LISTING AND FIGURE SHELLS

The following shells are provided in order to provide a framework for the display of data from this study. These shells may not be reflective of every aspect of this study but are intended to show the general layout of the Tables, Listings and Figures that will be included in the final clinical study report. Tables, Listings and Figures are numbered following the ICH structure. Table headers, variables names and footnotes will be modified as needed following data analyses. All descriptive and inferential statistical analyses will be performed using SAS® statistical software Version 9.4 or higher, unless otherwise noted.

TABLE, LISTING AND FIGURE SHELLS

01/12/2017 ■ Actavis LLC■ 

**T16.1.9.1 Summary of Discontinued Patients** 

| Patients | Test | Reference | Placebo | Total |
|---------------------|------|-----------|---------|-------|
| Randomized | XXX | XXX | XXX | XXX |
| Completed Study | XXX | XXX | XXX | XXX |
| Terminated Early | XXX | XXX | xxx | XXX |
| Lost to Follow-Up | XXX | XXX | xxx | XXX |
| Withdrew Consent | xxx | XXX | xxx | xxx |
| Randomized in Error | xxx | XXX | xxx | xxx |
| etc. | | | | |

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE  $^{\circledR}$  (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

**T16.1.9.2 Summary of Protocol Deviations** 

| | Test | Reference | Placebo | Total |
|-----------------------------------------|------|-----------|---------|-------|
| Total Patients with Protocol Deviations | XXX | XXX | xxx | XXX |
| Total Deviations | XXX | XXX | XXX | XXX |
| Outside Visit Window | XXX | XXX | XXX | XXX |
| Randomized in Error | XXX | XXX | XXX | XXX |
| Missed Visit | xxx | XXX | XXX | XXX |
| Restricted Medication | xxx | xxx | xxx | XXX |
| etc | XXX | xxx | xxx | XXX |
| Other | XXX | xxx | xxx | XXX |

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

**T16.1.9.3.1 Summary of Patients Excluded from Efficacy Analysis** 

01/12/2017 ■ Actavis LLC■ 

# **Ivermectin Cream 0.5%**

Protocol / Study No. 71691702

| | | Test | Reference | Placebo | Total |
|---|---|---|---|---|---|
| Randomized | Total | xxx | XXX | XXX | XXX |
| Safety Population | Total | xxx | XXX | xxx | xxx |
| Excluded from Safety | Total | xxx | XXX | XXX | XXX |
| | Not randomized or did not received study product | XXX | xxx | XXX | xxx |
| mITT Population | Total | XXX | XXX | xxx | XXX |
| Excluded from mITT | Total | XXX | XXX | xxx | xxx |
| | Did not dose | xxx | XXX | XXX | xxx |
| | etc. | | | | |
| PP Population | Total | xxx | XXX | xxx | xxx |
| Excluded from Excluded from PPP | Total | XXX | XXX | xxx | XXX |
| | Restricted Medication | xxx | xxx | xxx | XXX |
| | etc. | | | | |

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm


T16.1.9.3.2 Summary of Patients Included in Analysis Population by Study Center

| | | | | ] | PP | | | ml | TT | | | Safety | 7 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Site<br>No. | Name | Total<br>Randomized | Test | Reference | Placebo | Total | Test | Reference | Placebo | Total | Test | Reference | Placebo | Total |
| XXX | XXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

T16.1.9.4 Summary of Demographic Data and Baseline Characteristics (Safety Population)

| | | Test | Reference | Placebo | |
|---|---|---|---|---|---|
| | | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | P-value |
| Age (years) | n | XXX | XXX | xxx | x.xxxx |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | Median | XX.X | XX.X | XX.X | |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |
| Race | White | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | x.xxxx |
| | Black/African American | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Native Hawaiian or other Pacific Islander | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Asian | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | American Indian or Alaska Native | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | Other | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Gender | Female | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | x.xxxx |
| | Male | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |

N= number of patients in the specific treatment group; n= number of patient with data available; % is based on N

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE  $^{\circledR}$  (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

# T16.1.9.4 Summary of Demographic Data and Baseline Characteristics (Safety Population)

| | | Test | Reference | Placebo | |
|---|---|---|---|---|---|
| | | (N = xxx) | (N = xxx) | (N = xxx) | P-value |
| Ethnicity | Hispanic or Latino | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | x.xxxx |
| | Not Hispanic or Latino | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| Number of live lice | n | XXX | XXX | XXX | x.xxxx |
| | $Mean \pm SD$ | $xx.x \pm x.x$ | $\mathbf{x}\mathbf{x}.\mathbf{x} \pm \mathbf{x}\mathbf{x}.\mathbf{x}$ | $xx.x \pm xx.x$ | |
| | Median | XX.X | xx.x | xx.x | |
| | Range | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |

Note: N= number of patients in the specific treatment group; n= number of patient with data available; % is based on N

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE  $^{\circledR}$  (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

#### OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

Similar tables will be created for T16.1.9.5 and T16.1.9.6

T16.1.9.5 Summary of Demographic Data and Baseline Characteristics (modified Intent-to-Treat Population)

T16.1.9.6 Summary of Demographic Data and Baseline Characteristics (Per-Protocol Population)

01/12/2017 ■ Actavis LLC■ 

# T16.1.9.7 Summary of Analysis Results of Primary Efficacy Endpoint (Proportion of Index Patients with Treatment Successes between Treatment Groups)

| er-Protocol Populati | ion | | | |
|---|---|---|---|---|
| | | | Difference Between Treatments | |
| Number of | Number of Treatment | Proportion of Treatment | Difference (9/) | 90% CI Evaluation |
| | | | Difference (%) | 90% CI Evaluation |
| | | | XX.X | xx.x - xx.x |
| | • | Number of Treatment Patients (N) Successes (n) xxx xxx | Number of Proportion of Number of Treatment Treatment Patients (N) Successes (n) Successes (%) XXX XXX XXX XX.X | Number of Proportion of Number of Treatment Treatment Patients (N) Successes (n) Successes (%) Difference (%) XXX XXX XXX |

#### **Superiority: modified Intent-to-Treat Population**

| | | Number of | Proportion of | |
|-----------|--------------|---------------|---------------|---------|
| Treatment | Number of | Treatment | Treatment | |
| Group | Patients (N) | Successes (n) | Successes (%) | P-value |
| Placebo | XXX | XXX | XX.X | |
| Test | XXX | XXX | XX.X | x.xxxx |
| Reference | XXX | XXX | XX.X | X.XXXX |

Superiority of Active treatments over Placebo were tested using a two-sided Cochran-Mantel-Haenszel (CMH) test, stratified by clinical site, at the 5% significance level.

The superiority testing include patients in the mITT population using last observation carried forward (LOCF).

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm


# T16.1.9.8 Summary of Analysis Results of Secondary Efficacy Endpoint (Proportion of All Randomized Patients with Treatment Successes between Treatment Groups)

| <b>Equivalence:</b> P | Per-Protocol Populat | ion | | | |
|---|---|---|---|---|---|
| | | | | Difference Be | tween Treatments |
| | | Number of | Proportion of | | |
| Treatment | Number of | Treatment | Treatment | | |
| Group | Patients (N) | Successes (n) | Successes (%) | Difference (%) | 90% CI Evaluation |
| Test | xxx | xxx | XX.X | | |
| Reference | XXX | XXX | XX.X | XX.X | xx.x - xx.x |

#### **Superiority: modified Intent-to-Treat Population**

| | | Number of | Proportion of | |
|-----------|--------------|---------------|---------------|---------|
| Treatment | Number of | Treatment | Treatment | |
| Group | Patients (N) | Successes (n) | Successes (%) | P-value |
| Placebo | XXX | XXX | XX.X | |
| Test | XXX | XXX | XX.X | x.xxxx |
| Reference | XXX | XXX | XX.X | x.xxxx |

Superiority of Active treatments over Placebo were tested using a two-sided Cochran-Mantel-Haenszel(CMH) test, stratified by clinical site, at the 5% significance level.

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

T16.1.9.9 Overall Summary of Adverse Events (Safety Population)

| Description | Test | Reference | Placebo | Total |
|---|---|---|---|---|
| Patients Randomized | xxx | XXX | XXX | XXX |
| Patients with at least one AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Discontinued study drug due to above AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| AEs reported | XXX | XXX | xxx | XXX |
| Mild | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Moderate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Severe | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not Related | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Related | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Serious AE | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

# T16.1.9.10 Summary of Frequency of All Adverse Events by Body System (Safety Population)

| | | Test (N = xxx) | | | Reference $(N = xxx)$ | | $ Placebo \\ (N = xxx) $ | |
|---|---|---|---|---|---|---|---|---|
| Body System | MedDRA Term | Events | Patients | Events | Patients | Events | Patients | P-value |
| Patient with at least one AE | Total | XX | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) | x.xxxx |
| Ear and labyrinth<br>disorders | Ear pain | XX | xx (xx.x%) | XX | xx (xx.x%) | XX | xx (xx.x%) | x.xxxx |
| | etc. | | | | | | | |

etc.

Comparison of treatment groups is with respect to the number of patients with at least one occurrence of the AE.

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

T16.1.9.11 Summary of Frequency of All Adverse Events by Severity (Safety Population)

| | | | Test # Events (N=xx) | | | Reference # Events (N=xx) | | | Placebo<br># Events<br>(N=xx) | |
|---|---|---|---|---|---|---|---|---|---|---|
| <b>Body System</b> | MedDRA Term | Mild | Moderate | Severe | Mild | Moderate | Severe | Mild | Moderate | Severe |
| Total AEs | Total AEs | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ear and labyrinth disorders | Ear pain | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Hypoacusis | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx(xx.x%) | xx(xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

etc.

N = Total number of events in each treatment group; Percentage is based on total number of events.

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE  $^{\circledR}$  (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

T16.1.9.12 Summary of Frequency of All Adverse Events by Relationship (Safety Population)

| | | # E | Cest<br>events<br>=xx) | # E | erence<br>vents<br>=xx) | Placebo<br># Events<br>(N=xx) | |
|---|---|---|---|---|---|---|---|
| <b>Body System</b> | MedDRA Term | Related | Not Related | Related | Not Related | Related | Not Related |
| Total AEs | Total AEs | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ear and labyrinth | Ear pain | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| disorders | Hypoacusis | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | etc. | | | | | | |

etc.

N = Total number of events in each treatment group; Percentage is based on total number of events.

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

# T16.1.9.13 Summary of Frequency of Serious Adverse Events (Safety Population)

| | | Test | Reference | Placebo |
|---|---|---|---|---|
| Body System | MedDRA Term | # Events | # Events | # Events |
| Injury, poisoning and procedural complications | Alcohol poisoning | XX | XX | XX |

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 
T16.1.9.14 Summary of Frequency of Application Site Reaction (Safety Population)

| Signs and | | | Placebo | Test | Reference |
|---|---|---|---|---|---|
| Symptoms | Visit | Statistic | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N}=\mathbf{x}\mathbf{x})$ |
| Edema | Visit 1 | Absent | xxx (x.x%) | xxx (x.x%) | xxx (x.x%) |
| | | Mild | xxx (x.x%) | xxx (x.x%) | xxx (x.x%) |
| | | Moderate | xxx (x.x%) | xxx (x.x%) | xxx (x.x%) |
| | | Severe | xxx (x.x%) | xxx (x.x%) | xxx (x.x%) |
| | Visit 2 | | | | |
| | Visit 3 | | | | |
| | Visit 4 | | | | |

Erythema

Excoriation

Pain

Pruritus

Pyoderma

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

# T16.1.9.15 Summary of Vital Signs (Safety Population)

| Vital Signs | Visit | Statistic | Test (N = xxx) | Reference $(N = xxx)$ | $\begin{aligned} & \text{Placebo} \\ & (\mathbf{N} = \mathbf{x} \mathbf{x} \mathbf{x}) \end{aligned}$ |
|---|---|---|---|---|---|
| Systolic Blood Pressure (mmHg) | Visit 1 | n | XXX | XXX | XXX |
| | | $Mean \pm SD$ | $xxx.x \pm xxx.x$ | $xxx.x \pm xxx.x$ | $xxx.x \pm xxx.x$ |
| | | Median | XXX.X | xxx.x | xxx.x |
| | | Range | xxx.x - xxx.x | xxx.x - xxx.x | xxx.x - xxx.x |
| | Visit 2 | | | | |
| | Visit 3 | | | | |
| | Visit 4 | | | | |

Diastolic Blood Pressure (mmHg)

Heart Rate (beats/min)

Respiration Rate (breaths/min)

Temperature (F)

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE  $^{\circledR}$  (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

#### STATISTICAL ANALYSIS PLAN

#### **Ivermectin Cream 0.5%**

Protocol / Study No. 71691702


T16.1.9.16

# (Safety Population)

| Visit | Test (N = xxx) | Reference<br>(N = xxx) | Placebo<br>(N = xxx) |
|-------|----------------|------------------------|----------------------|
| | xxx (x.x%) | xxx (x.x%) | xxx (x.x%) |
| | xxx (x.x%) | xxx (x.x%) | xxx (x.x%) |

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm


T16.1.9.17

# (Safety Population)

| Test (N = xxx) | Reference $(N = xxx)$ | Placebo<br>(N = xxx) |
|----------------|-----------------------|----------------------|
| xxx (x.x%) | xxx (x.x%) | xxx (x.x%) |

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

Re-infestation is defined as treatment success at Visit 2 and treatment failure at either Visit 3 or 4, or treatment success at Visits 2 and 3 and treatment failure at Visit 4.

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

## L16.2.1 Listing of Discontinued Patients

| Treatment | Patient | Discontinuation | scontinuation |
|-----------|------------|-------------------|---------------|
| Group | Number | Reason | Population |
| Test | xxx-xxx-xx | Withdrew Consent | mITT |
| | XXX-XXX-XX | Lost to Follow-up | Safety |

Reference

Placebo

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

#### L16.2.2 Listing of Protocol Deviations

| Treatment | Patient | | |
|-----------|------------|-----------------------------------|------------|
| Group | Number | <b>Protocol Deviation Summary</b> | Population |
| Test | XXX-XXX-XX | Outside Visit Window | Safety |

Reference

Placebo

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

#### L16.2.3.1 Listing of Patients Excluded from the Per-Protocol Population

| Treatment<br>Group | Patient<br>Number | Exclusion<br>Reason |
|--------------------|-------------------|-------------------------------------|
| Test | XXX-XXX-XX | Patient did not meet IE criterion. |
| | XXX-XXX-XX | Patient took prohibited medications |

Reference

Placebo

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

#### L16.2.3.2 Listing of Patients Excluded from the Modified Intent-to-Treat Population

| Treatment<br>Group | Patient<br>Number | Exclusion<br>Reason |
|---|---|---|
| Test | xxx-xxx-xx | Patient did not have at least one post-randomization evaluation |
| | xxx-xxx-xx | Patient did not have at least one post-randomization evaluation |

Reference

Placebo

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

## L16.2.4.1 Listing of Demographic Data

| Treatment | Patient | | | | |
|---|---|---|---|---|---|
| Group | Number | Age | Gender | Ethnicity | Race |
| Test | xxx-xxx-xx | 30 | Female | Not Hispanic or Latino | Black or African American |

Reference

Placebo

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE  $^{\circledR}$  (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

# L16.2.4.2 Listing of Medical History

| Treatment | reatment Patient Diagnosis or Surgical | | | | | |
|---|---|---|---|---|---|---|
| Group | Number | System | Procedure | Start Date | <b>End Date</b> | Ongoing |
| Test | XXX-XXX-XX | Gynecologic | Menopause | 2003 | 2003 | |

Reference

Placebo

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

# L16.2.4.3 Listing of Concomitant Medications

| Treatment | Patient | | TX | | | | Start/End | |
|---|---|---|---|---|---|---|---|---|
| Group | Number | Medication | Area | Dosage | Frequency | Route | Date | Indication |
| Test | xxx-xxx-xx | LISINOPRIL | Yes | 20 MG | QD | РО | yyyy-mm-dd/ | HYPERTENSION |
| | | | | | | | yyyy-mm-dd | |

Reference

Placebo

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

# L16.2.5 Listing of Visit Date Information

| Treatment | Patient | Informed Consent | | | | Visit 4 or |
|---|---|---|---|---|---|---|
| Group | Number | Date | Visit 1 | Visit 2 | Visit 3 | Discontinuation |
| Test | xxx-xxx-xx | yyyy-mm-dd | yyyy-mm-dd | yyyy-mm-dd | yyyy-mm-dd | yyyy-mm-dd |

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

# L16.2.6 Listing of Louse Examination Results

| Treatment<br>Group | Patient<br>Number | Visit | Were Live Head<br>Lice Present? | Number of Live<br>Head Lice | Treatment<br>Success | Duration of Louse<br>Examination<br>(minutes) |
|---|---|---|---|---|---|---|
| Test | xxx-xxx-xx | Visit 1 | Yes | 6 | | XX |
| | | Visit 2 | Yes | 5 | | XX |
| | | Visit 3 | Yes | 2 | | XX |
| | | Visit 4 | No | 0 | Yes | XX |
| | XXX-XXX-XX | Visit 1 | Yes | 6 | | XX |
| | | Visit 2 | Yes | 5 | | XX |
| | | Visit 3 | Yes | 2 | | XX |
| | | Visit 4 | Yes | 2 | No | XX |
| | etc | | | | | |

Reference Placebo

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

#### L16.2.7.1 Listing of Adverse Events by Treatment Group

| Treatment group | Patient<br>Number | Body System/<br>MedDRA Term/<br>AE Term | TX<br>Area | Start /End<br>Date | Severity | Relationship<br>to Study<br>Drug | Outcome | Action Taken with<br>Study Drug/<br>Other Action<br>Taken | SAE? |
|---|---|---|---|---|---|---|---|---|---|
| Test | XXX-XXX-XX | Nervous system disorders/ headache/ | No | yyyy-mm-dd / | Mild | Not Related | Recovered | Drug withdrawn/ None | No |
| | | Headache | | yyyy-mm-dd | | | | | |

Reference

Placebo

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

# L16.2.7.2 Listing of Application Site Reactions

| Treatment<br>Group | Patient<br>Number | Visit | Edema | Erythema | Excoriation | Pain | Pruritus | Pyoderma |
|---|---|---|---|---|---|---|---|---|
| Test | xxx-xxx-xx | Visit 1 | 0 | 0 | 0 | 1 | 0 | 0 |
| | | Visit 2 | 0 | 1 | 0 | 0 | 0 | 0 |
| | | Visit 3 | 0 | 0 | 0 | 1 | 0 | 0 |
| | | Visit 4 | 0 | 0 | 0 | 1 | 0 | 0 |

Reference

Placebo

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

# L16.2.8.1 Listing of Pregnancy Test Results

| Treatment | Patient | | | | Visit 4 or |
|-----------|------------|----------|----------|----------|-----------------|
| Group | Number | Visit 1 | Visit 2 | Visit 3 | Discontinuation |
| Test | XXX-XXX-XX | Negative | Negative | Negative | Negative |

Reference

Placebo

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 

# L16.2.8.2 Listing of Vital Signs

| Treatment | Patient | | Systolic BP | Diastolic BP | Pulse Rate | Respiration Rate | Temperature |
|---|---|---|---|---|---|---|---|
| Group | Number | Visit | (mmHg) | (mmHg) | (beats/min ) | (breaths/min) | <b>(F)</b> |
| Test | xxx-xxx-xx | Visit 1 | 120 | 70 | 84 | 18 | 98.6 |
| | | Visit 2 | 140 | 80 | 74 | 18 | 97 |
| | | Visit 3 | 120 | 70 | 84 | 18 | 98.6 |
| | | Visit 4 | 140 | 80 | 74 | 18 | 97 |

Reference

Placebo

Test: Ivermectin Lotion, 0.5% (Actavis Laboratories UT, Inc.)

Reference: SKLICE® (ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC)

Placebo: Placebo (vehicle) lotion (Actavis Laboratories UT, Inc.)

OUTPUT: L:\DEV\917\71691702\SAS\OUT\XXXX

Created on: ddmmmyy hh:mm Page 1 of N

01/12/2017 ■ Actavis LLC■ 